CLINICAL TRIAL: NCT06831747
Title: MiniLap Vs Standard Laparoscopy in Prophylactic Bilateral Salpingo-Oophorectomy in BRCA-Mutated Patients: a Randomized Controlled Trial
Brief Title: MiniLap Vs Standard Laparoscopy in Prophylactic Bilateral Salpingo-oophorectomy in BRCA-Mutated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Stefano Restaino, Doctor, Azienda Sanitaria-Universitaria Integrata di Udine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0022677
Record Dates: First submitted 2025-01-19; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: BRCA Mutation
Keywords: Laparoscopy; BRCA mutations; Salpingo-Oophorectomy; MiniLap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Standard laparoscopy (Active Comparator): Bilateral salpingo-oophorectomy performed with standard laparoscopy
  Interventions: Procedure: Bilateral salpingo-oophorectomy - S-LPS
- B: MiniLap (Experimental): Bilateral salpingo-oophorectomy performed with MiniLap
  Interventions: Procedure: Bilateral salpingo-oophorectomy - PSS

INTERVENTIONS:
Procedure: Bilateral salpingo-oophorectomy - S-LPS — In standard laparoscopy (S-LPS), the initial laparoscopic access was performed at the umbilical level using open laparoscopy (Hasson technique). The subsequent accesses were carried out in the right and left iliac fossa. In the S-LPS, these accesses are performed using a 5mm trocars. Finally, a 5mm ancillary trocar was placed in the suprapubic region to use instruments such as bipolar forceps, irrigators, and scissors. The subsequent surgical steps were identical for both techniques.
  Arms: A: Standard laparoscopy
Procedure: Bilateral salpingo-oophorectomy - PSS — In the MiniLap® Percutaneous Surgical System (PSS), the initial laparoscopic access was performed at the umbilical level using open laparoscopy (Hasson technique). The subsequent two accesses were carried out in the right and left iliac fossa. These latter accesses are directly performed using MiniLap® with a 2.4mm incision. Finally, a 5mm ancillary trocar was placed in the suprapubic region to use instruments such as bipolar forceps, irrigators, and scissors. The subsequent surgical steps were identical for both techniques.
  Arms: B: MiniLap

SUMMARY:
The study hypothesis is that surgical treatment performed with MiniLap results in reduced postoperative pain in a population of patients undergoing prophylactic laparoscopic adnexal surgery. The primary objectives are to assess differences in operative duration, intraoperative blood loss, and postoperative complications in patients undergoing bilateral laparoscopic adnexectomy performed with standard laparoscopy versus MiniLap. The secondary objectives of this study are to compare postoperative pain and patient satisfaction with aesthetic outcomes.

Patients with BRCA 1/2 mutations undergoing prophylactic surgery will be assigned to either MiniLap or standard laparoscopic treatment based on randomization. Subsequently, the necessary study data will be collected using the hospital's electronic management system and medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing prophylactic bilateral adnexectomy via laparoscopic surgery.
* Patients with a germline mutation in the BRCA1/2 gene.

Exclusion Criteria:

* Patients who underwent additional surgery during the adnexectomy procedure.
* Patients in whom an intraoperative frozen section is required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative outcomes: operative time (minutes), intraoperative blood loss (mL), postoperative complications (clavien dindo classification) | From enrollment to 30 days postoperatively
  The primary objectives are to assess differences in:
  operative time (minutes), intraoperative blood loss (mL), postoperative complications (clavien dindo classification) in patients undergoing bilateral laparoscopic adnexectomy performed with standard laparoscopy versus MiniLap.

SECONDARY OUTCOMES:
Pain (Visual Analog Score) | From enrollment to 2 days postoperatively.
  The secondary objective of this study is to compare postoperative pain (VAS 0-10; higher scores mean worse)
Cosmetic results (Visual Analog Score) | From enrollment to 60 days postoperatively.
  The secondary objective of this study is to compare patient satisfaction with aesthetic outcomes using a VAS scale (0-10, with higher scores indicating greater satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Maternal and Child Health, Obstetrics and Gynecology Clinic, University Hospital of Udine, Udine, Udine, Italy